CLINICAL TRIAL: NCT02794532
Title: Pre-oxygenation With High-flow Nasal Cannula in Comparison to Standard in Adults During Rapid Sequence Induction Anesthesia- a Prospective Randomized Non-blinded Clinical Trial
Brief Title: PreOxygenation In RSI Anesthesia
Acronym: PRIOR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska University Hospital (Other)
Responsible Party: Principal Investigator, Malin Jonsson Fagerlund, Associate Professor, senior Consultant, Karolinska University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PRIOR
Record Dates: First submitted 2016-05-11; First posted 2016-06-09 (Estimated); Last update posted 2017-12-19 (Actual); Status verified 2017-12

CONDITIONS: Anesthesia; Oxygen

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Pre oxygenation with 100% oxygen via tight fitting mask (No Intervention): Pre Oxygenation will be done using a tight mask
- Pre oxygenation with 100% oxygen in high-flow nasal cannula (Experimental): Pre Oxygenation will be done using high-flow nasal canula
  Interventions: Procedure: High-flow nasal cannula

INTERVENTIONS:
Procedure: High-flow nasal cannula — Oxygenation will be done via a high-flow nasal cannula
  Arms: Pre oxygenation with 100% oxygen in high-flow nasal cannula

SUMMARY:
Pre-oxygenation with high-flow nasal cannula oxygen has been evaluated in a limited number of studies and seems to be better than traditional preoxygenation with a tight fitting mask. Oxygenation with high-flow nasal cannula in apnea demonstrates that this could be done safely for up to 25 mins with preserved saturation. Based on this, the investigators want to evaluate whether this novel concept of preoxygenation can prolong the time to desaturation in emergency anesthesia while securing a possibly difficult airway. This may reduce the number of hypoxic events during intubation. This novel concept has already been tested in clinical practice in certain cases but not during rapid sequence induction for acute surgery.

Objectives and Purpose The general purpose of this project is to compare a new preoxygenation technique based on humidified oxygen in a high-flow nasal cannula with traditional preoxygenation with a tight fitting mask during rapid sequence induction intubation with focus on gas exchange.

DETAILED DESCRIPTION:
Pre-oxygenation with high-flow nasal cannula with 100% oxygen has been evaluated in a limited number of studies and seems to be equal or better than traditional preoxygenation with tight fitting mask. Apneic oxygenation with high-flow nasal cannula in apnea demonstrates that this could safely be don up to 25 minutes. Based on this, we can to evaluate whether this novel concept of preoxygenation can prolong the time before desaturation in emergency anesthesia and a difficult airway situation. This could ultimately reduce the number of damage to the airway and hypoxic injuries. This novel concept is already tested in clinical practice in certain cases and we strongly believe that a scientific evaluation of this approach is needed before a broad implementation.

The patients will undergo regular pre-anesthetic evaluation and will be then be asked to participate in the study. Oral and written information will be given. A consent form will be signed.

The patients will be randomized to either traditional preoxygenation or preoxygenation with high-flow nasal cannula (HFNC) oxygen.

On arrival in the operating room standard patient monitoring will be applied (ECG, pulse oximetry, non-invasive blood pressure) and preparation for anesthesia induction will be done with the patients placed with a slightly elevated head, approximately 25º. Peripheral oxygen saturation (SpO2) will be noted when breathing room air. If an arterial line is planned this will be put in place before pre-oxygenation and a blood sample will be drawn when breathing room air Preoxygenation will hereafter take place either the traditional way or with a HFNC. The traditional preoxygenation consists of breathing 100% oxygen via a tight-fitting non-rebreathing facial mask with a fresh gas flow of ≥10 L/min of for ≥ 3 minutes. HFNC pre-oxygenation consists of application of nasal cannulae (Optiflow TM, Fisher & Paykel Healthcare, Auckland, New Zealand) in the nostrils and the patients will receive 40L/min of heated and humidified 100% oxygen for ≥ 3 minutes.

After induction of anesthesia with RSI the airways will be kept open by manual adjustment by the anesthesiologist until intubation regardless of pre-oxygenation technique. During the laryngoscopy and intubation 70L/min of humidified 100% oxygen will be administered continuously by the nasal cannula left in place if HFNC oxygen is used.

Endtidal carbon dioxide (ETCO2) will be noted before the start of pre-oxygenation and on the first breath after intubation. If an arterial line is in place blood gas samples will be taken before the start of pre-oxygenation (breathing room air) and when the endotracheal tube is in place.

Output data:

* SpO2 breathing room air, at end of pre-oxygenation and one minute after intubation
* ETCO2 before pre-oxygenation and at first breath after intubation
* Time to intubation (measured from start of laryngoscopy to when ET tube correctly in place)
* Total time of high flow nasal cannula oxygen /traditional pre-oxygenation delivered
* Blood pressure
* Heart rate
* ASA classification level
* Smoker/non-smoker
* BMI
* Preoperative presence of lung condition (eg. chronic obstructive pulmonary disease (COPD), asthma) yes/no
* Preoperative oxygen therapy
* Known/treated obstructive sleep apnea (OSA) yes/no
* Type of surgery: abdominal yes/no
* Duration of surgery, hours
* Mallampati grade, thyromental distance, mouth opening and neck movement.
* Cormack & Lehane grade
* Number of attempts to intubate
* Use of bougie during intubation yes/no
* Cricoid pressure used yes/no
* Clinical suspicion of aspiration on intubation
* Subjective experience of the pre oxygenation measured on a Visual Analogue Scale

Disruption criteria The patient doesn´t tolerate pre-oxygenation the way it is planned according to randomization.

Statistics This is a randomized controlled study evaluating a novel concept and comparing it to a traditional technique. Continuous data will be presented as mean ± SD or 95% CI and categorical data as median and range. We will analyze the data using Prism 6.0 (GraphPad) or SPSS 24 (IBM). We do not know the primary outcome parameters (lowest saturation within 1 min after intubation), but with an estimation based partly on a previous study (Wimasalena et al. Ann Emerg Med 2015) we assume that the lowest saturation in the control group will be 93% and 95% in the treatment group with a SD of 3%. Using a type I error of 5% and type II error of 20% (power 80%) a sample size of 70 patients in each group was calculated. To allow for missed data and drop-outs we plan to include 100+100 patients (total of 200 patients). After inclusion of 80 patients an interim analysis will be performed for the primary outcome. A non-paired t-test will be performed to analyse the primary outcome.

ELIGIBILITY:
Inclusion Criteria:

1. Adult, >18 years old
2. Emergency intubation where RSI is indicated
3. Capable of understanding the study information and signing the written consent.
4. Need for non-invasive ventilation

Exclusion Criteria:

1. BMI >35
2. Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2016-06-01 (Actual); Primary Completion 2017-06-01 (Actual); Study Completion 2017-10-01 (Actual)

PRIMARY OUTCOMES:
Lowest peripheral oxygen saturation from induction of anaesthesia to 1 minute after tracheal intubation | One minute after tracheal intubation
  Peripheral oxygen saturation will be measured. The lowest value from start of anesthesia until up to 1 minute after tracheal intubation is the primary outcome measure.

SECONDARY OUTCOMES:
Change in level of oxygen saturation during high flow nasal cannula oxygenation compared with traditional pre-oxygenation from time to first anesthetic drug given to 1 minute after intubation. | One minute after tracheal intubation
Number of patients with desaturation below 93 % with high flow nasal cannula oxygenation compared with traditional pre-oxygenation? | One minute after tracheal intubation
Level of end tidal carbon dioxide in the first breath after intubation with high flow nasal cannula oxygenation compared with traditional pre-oxygenation? | First breath after endotracheal intubation
Degree of discomfort with pre oxygenation for the patient | The assessment will be done at the postoperative unit
  The degree of discomfort for the patients will be assessed with a visual analogue scale ranging from 0- 10, where 10 is maximal discomfort

CONTACTS AND LOCATIONS:
Overall Officials: Malin Jonsson Fagerlund, Principal Investigator — Karolinska University Hospital and Karolinska Institutet

IPD SHARING:
Plan to Share IPD: Undecided